CLINICAL TRIAL: NCT05019378
Title: Evaluation of the Autologous Stromal Vascular Fraction Therapy for Knee Osteoarthritis
Brief Title: SVF Therapy for Human Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhongnanzxx
Record Dates: First submitted 2021-08-10; First posted 2021-08-24 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Knee Osteoarthritis
Keywords: Cartilage Defect; Cartilage Regeneration
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous SVF treatment (Experimental): Three milliliter of cell suspension injection containing 1.0E8 SVF cells into the knee joint
  Interventions: Procedure: SVF treatment
- Placebo group (No Intervention): No treatment

INTERVENTIONS:
Procedure: SVF treatment — autologous SVF (10E8 cells)
  Arms: autologous SVF treatment

SUMMARY:
The purpose of the study is to asses the safety and efficacy of SVF for treatment of knee osteoarthritis, and establish a novel method to provide 3D MRI imaging for human knee cartilage to qualitatively and quantitatively evaluate cartilage regeneration.

DETAILED DESCRIPTION:
Study participants voluntarily provided written informed consent to participate in the study. The two knees of each patient were randomly assigned to autologous SVF treatment group or non-treatment control group. The patients were evaluated every 4 weeks for safety and efficacy of autologous SVF therapy for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Knee Osteoarthritis
* Articular cartilage defect grades I/II of both knee

Exclusion Criteria:

* autoimmune or inflammatory arthritis
* serious medical disorders

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Radiologic evaluation of knee articular cartilage Volume | Change from Baseline articular cartilage Volume at 12 weeks
  The Volume (cubic millimeter) of knee articular cartilage are measured.
Radiologic evaluation of knee articular cartilage Volume | Change from Baseline articular cartilage Volume at 24 weeks
  The Volume (cubic millimeter) of knee articular cartilage are measured.
Radiologic evaluation of knee articular cartilage Area | Change from Baseline articular cartilage Area at 12 weeks
  The Area (square millimeter) of knee articular cartilage are measured.
Radiologic evaluation of knee articular cartilage Area | Change from Baseline articular cartilage Area at 24 weeks
  The Area (square millimeter) of knee articular cartilage are measured.
Radiologic evaluation of knee articular cartilage Thickness | Change from Baseline articular cartilage Thickness at 12 weeks
  The Thickness (millimeter) of knee articular cartilage are measured.
Radiologic evaluation of knee articular cartilage Thickness | Change from Baseline articular cartilage Thickness at 24 weeks
  The Thickness (millimeter) of knee articular cartilage are measured.
Knee pain evaluation and functional evaluation (the Western Ontario and McMaster University arthritis index [WOMAC]) | Change from Baseline WOMAC arthritis index score at 12 weeks.
  Knee pain and functional mobility were assessed using WOMAC arthritis index patient questionnaire including 24 parameters for pain, stiffness and physical function. The values ranging from 0 (minimum) to 240 (maximum) and the lower scores mean a better outcome.
Knee pain evaluation and functional evaluation (the Western Ontario and McMaster University arthritis index [WOMAC]) | Change from Baseline WOMAC arthritis index score at 24 weeks.
  Knee pain and functional mobility were assessed using WOMAC arthritis index patient questionnaire including 24 parameters for pain, stiffness and physical function. The values ranging from 0 (minimum) to 240 (maximum) and the lower scores mean a better outcome.
Knee pain evaluation and functional evaluation (The Lysholm Knee Scoring Scale) | Change from Baseline Lysholm Knee Scale score at 12 weeks.
  The Lysholm Knee Scoring Scale questionnaire has been designed to evaluate how patients' knee pain has affected their ability to manage everyday life. The values ranging from 0 (minimum) to 100 (maximum) and the higher scores mean a better outcome.
Knee pain evaluation and functional evaluation (The Lysholm Knee Scale) | Change from Baseline Lysholm Knee Scale score at 24 weeks.
  The Lysholm Knee Scoring Scale questionnaire has been designed to evaluate how patients' knee pain has affected their ability to manage everyday life. The values ranging from 0 (minimum) to 100 (maximum) and the higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Xiao Zheng, MD, Principal Investigator — Wuhan University; Lin Cai, MD, Study Director — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: starting 6 months after publication